CLINICAL TRIAL: NCT02571582
Title: Predictors of Mortality in Patients With Advanced Lung Disease in Home Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Vinícius Pafume de Oliveira, Physiotherapist, Federal University of Uberlandia
Other Study IDs: Study of Advanced Lung Disease
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Obstructive Pulmonary Disease and Allied Conditions
Keywords: Predictors of mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients died: All patients underwent extensive evaluation:
  - Body composition, Diabetes; dyslipidemia, hemoconcentration, hypertension, exercise capacity: 6-Minute Walk test procedure, renal function, inflammatory markers, cause and place of death, time tracking concentrator, quality of life and pulmonary Function.
- living patients: All patients underwent extensive evaluation:
  - Body composition, Diabetes; dyslipidemia, hemoconcentration, hypertension, exercise capacity: 6-Minute Walk test procedure, renal function, inflammatory markers, cause and place of death, time tracking concentrator, quality of life and pulmonary Function.

SUMMARY:
Advanced Pulmonary Disease (PAD) is a condition that affects countless individuals around the world. Patients are often functionally very limited, with premature death, which is due to the disease itself or its complications. Currently, there are numerous monitoring centers of these patients to increase survival, reduce costs and humanize care in these patients.

DETAILED DESCRIPTION:
The advanced chronic lung disease (PAD) is characterized by the development of several structural abnormalities, and pulmonary and systemic functional with low potential for reversibility, in spite of the treatment. It is defined DPA whole lung non-neoplastic chronic in its final phase. Most people with DPA consists of elderly people who have lung function and quite compromised gas exchange. These conditions determine chronically limitations in activities of daily living, negative impact on mental and social state, frequent exacerbations of the disease and numerous hospitalizations, recognized risk factors for increased morbidity and mortality (MACHADO, 2006).

Clinically, patients with APD may have one or more of the following signs and symptoms: dyspnea; cough; intolerance efforts; hypoxemia and / or hypercapnia; malnutrition and / or cachexia; anxiety and / or depression (BTS 2004).

According Garden 2004, the DPA affects millions of people worldwide and it is estimated that in Brazil there are two million individuals with APD. The most prevalent lung diseases, which in the final stage, fall under the DPA definition are classified as obstructive, restrictive, vascular and hypoventilation syndromes. Obstructive chronic respiratory insufficiency are part individuals with COPD, bronchiectasis and other bronchiolitis. Already restrictive covers patients with interticiais diseases and neuromuscular diseases. And the pulmonary vascular diseases fit patients with primary pulmonary hypertension and secondary and chronic pulmonary thromboembolism (MACHADO, 2006; PAUL, 2005).

Within the restrictive diseases with high prevalence we find the interticiais diseases are heterogeneous disorders, grouped according to clinical, radiological and functional similar. In the group of conditions that account for the majority of advanced pulmonary diseases are idiopathic pulmonary fibrosis, hypersensitivity pneumonitis and sarcoidosis. The etiology is unknown in many situations; and any known causes that stand out are the tobacco-related diseases (Guidelines interticiais lung diseases, 2012).

Vascular diseases also fits in advanced lung disease and presents significant pulmonary and systemic changes in patients. Before insulting stimuli of different nature, the pulmonary vessels undergo changes, known as pathological remodeling of the circulation. The vessel is tougher and reactive, causing pulmonary vascular diseases. Morphologic lesions in the arterial tree leads to local changes in the pattern of blood flow, that flow slowly added to the changes detected in the endothelial surface and abnormalities of the coagulation system proteins provide local thrombus formation. Pulmonary hypertension is a pathological condition that is present when the mean pulmonary artery pressure above 25 mmHg (CONSENSUS, 2009).

The alveolar hypoventilation is the major injury to the respiratory function by obesity. The concept of alveolar hypoventilation reflects the incompetence of the respiratory system to eliminate carbon dioxide in the same proportion that reaches the lungs. Implies, therefore, the presence hypercapnia (PaCO2> 45 mm Hg) accompanied by equivalent degree of hypoxemia (low PaO 2). Alveolar hypoventilation syndrome-obesity is defined as chronic alveolar hypoventilation in obese patients (body mass index greater than 30 kg / m2), without any other respiratory disease to justify the disorder of gas exchange. Palliative treatment consists in controlling chronic hypoventilation and hypoxemia and resolute treatment is to combat obesity (SILVA, GA 2006).

Among the obstructive diseases of major relevance are bronchiectasis and COPD. Bronchiectasis refers to the dilatation of the bronchi and irreversible distortion due to the destruction of the elastic and muscle component of its wall. It can be congenital or acquired. To purchase no need to aggression by an infection and disability in hygiene bronchial secretions. The patient has a cough, possibly with episodes of hemoptysis (GARDEN, 2004).

COPD is a preventable and treatable respiratory disease characterized by the presence of chronic airflow obstruction that is not fully reversible. The airflow obstruction is usually progressive and associated with an abnormal inflammatory response of the lungs to inhaled particles or toxic gases. Although COPD affects the lungs, it also produces significant systemic consequences that contribute to disease severity (GOLD - Global Obstructive Lung Disease, 2013).

The ODP is considered a non-pharmacological treatment critical for patients with chronic respiratory insufficiency. Maintaining low and stable level of oxygen in blood is of great importance for the organic homeostasis. Oxygen supplementation improves survival of patients with chronic hypoxemia and your prescription is recommended in the consensus on the subject. The main benefits of oxygen to the body are the decline in ventilatory work and improves the cardiovascular and muscular functions (Machado, 2006).

Classical studies have found that the use of ODP for more than 15 h / day in patients with chronic respiratory diseases increases survival in patients with severe hypoxemia (Lancet, 1981; Ann Intern Med, 1980...). The use of oxygen is indicated in patients with (as GOLD - Global Obstructive Lung Disease, 2013):

* PaO2 mmHg or SpO2 ≤ 55 ≤ 88, with or without hypercapnia confirmed two times over a period of 3 weeks, or
* = 55 to 60 mmHg PaO2 or SaO2 = 89%, with evidence of pulmonary hypertension, or polycythemia (hematocrit> 55%) The number of patients who require ODP is increasing every year. This type of therapy is being used more frequently in order to reduce morbidity and mortality and improve the quality of life of patients. This practice allows you to optimize the occupation of the beds, reduce the length and the number of hospitalizations and thus reduce hospital costs (Tanni, S. E et al 2007).

Two large studies have evaluated the benefits of ODP. The first study conducted by the Medical Research Concil compared the use of oxygen for 15h / d X 0 h / d, showing improved survival in those patients who regularly used oxygen. The second study, the Nocturnal Oxygen Therapy Trial, compared the use of 24h / d with 12h / d, showing improved survival in those patients who used oxygen for longer (Nocturnal Oxygen Therapy Trial Group, 1980).

The DPA's are an important public health problem in the world. Many people suffering from these diseases for years and die prematurely from the disease itself or its complications. The DPA, particularly COPD, are classified as a major cause of morbidity and mortality worldwide and results in an economic and social impact is substantial and growing, the debt is having a major highlight in the medical field in recent years (Gold, 2013).

Thus this work will identify the predictors of mortality in patients with DPA in ODP and help professionals and public and private policy health directly linked to treat these patients, to optimize the clinical management, helping improve the treatment of these patients, increasing life expectancy, reducing costs and improving the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

Advanced Pulmonary disease using home oxygen therapy;

• Have a diagnosis of chronic hypoxemia proven by blood gas analysis on room air PaO 2 ≤ 55 mm Hg or SaO2 ≤ 88; or PaO2 between 55 and 60 mmHg or SaO2 between 89 and 90%, with evidence of pulmonary hypertension, or polycythemia (hematocrit> 55%) as GOLD - Global Obstructive Lung Disease, 2015;

Exclusion Criteria:

No records found Patients who failed to perform the periodic reviews established by the team responsible

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients with established diagnosis of advanced lung disease that makes / made long home Oxygen use which were accompanied or followed at Oxygen Therapy Clinic of the Federal University of Uberlândia (UFU) by the Home Care Program (PAD), from 2009 to 2015. The sampling is for convenience.
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determine the predictors of mortality in patients with DPA in use of ODP | 6 years
  Evaluate the results of evaluations carried out in patients who died and had advanced lung disease diagnosis in use of home oxygen, compared to patients who did not die and the normal population

SECONDARY OUTCOMES:
Assess adherence to the use of home oxygen and its relation to the survival of these patients; | 6 years
  Assess the amount of oxygen that was used by patients during treatment indication and measurement of variable
To evaluate the influence of quality of life in patient survival; | 6 years
  Measure the quality of life of these patients and compared with the normal population and patients who died and had survival for longer period

OTHER OUTCOMES:
Identify the causes of mortality of these patients. | 6 years
  Search the causes of death of these patients and the place to compare with the current epidemiology and relate to the main disease

CONTACTS AND LOCATIONS:
Overall Officials: Vinícius Oliveira, Pafume, Principal Investigator — Federal Principal Investigator

REFERENCES:
- [Result] Holmes DR Jr, Dehmer GJ, Kaul S, Leifer D, O'Gara PT, Stein CM. ACCF/AHA clopidogrel clinical alert: approaches to the FDA "boxed warning": a report of the American College of Cardiology Foundation Task Force on clinical expert consensus documents and the American Heart Association endorsed by the Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. J Am Coll Cardiol. 2010 Jul 20;56(4):321-41. doi: 10.1016/j.jacc.2010.05.013. No abstract available. PMID 20633831
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Tomioka K, Iwamoto J, Saeki K, Okamoto N. Reliability and validity of the International Physical Activity Questionnaire (IPAQ) in elderly adults: the Fujiwara-kyo Study. J Epidemiol. 2011;21(6):459-65. doi: 10.2188/jea.je20110003. Epub 2011 Sep 24. PMID 21946625
- [Result] Shah T, Jagpal S, Beckford R. Long-acting bronchodilators in patients with chronic obstructive pulmonary disease: still more to know. Ann Am Thorac Soc. 2014 Nov;11(9):1504. doi: 10.1513/AnnalsATS.201409-439LE. No abstract available. PMID 25423005
- [Result] Kim AL, Kwon JC, Park I, Kim JN, Kim JM, Jeong BN, Yu SK, Lee BK, Kim YJ. Reference equations for the six-minute walk distance in healthy korean adults, aged 22-59 years. Tuberc Respir Dis (Seoul). 2014 Jun;76(6):269-75. doi: 10.4046/trd.2014.76.6.269. Epub 2014 Jun 28. PMID 25024720
- [Result] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Result] Velloso M, Jardim JR. Functionality of patients with chronic obstructive pulmonary disease: energy conservation techniques. J Bras Pneumol. 2006 Nov-Dec;32(6):580-6. doi: 10.1590/s1806-37132006000600017. English, Portuguese. PMID 17435910
- See also: The Global Initiative for Chronic Obstructive Lung Disease (GOLD) works with health care professionals and public health officials to raise awareness of Chronic Obstructive Pulmonary Disease (COPD) and to improve prevention and treatment of this lung di — http://www.goldcopd.com/